CLINICAL TRIAL: NCT04076293
Title: A First-in-Human, Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM15912(Sonefpeglutide) in Healthy Korean Subjects
Brief Title: Single Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM15912(Sonefpeglutide) in Healthy Korean Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hanmi Pharmaceutical Company Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HM-GLP2-101
Record Dates: First submitted 2019-08-26; First posted 2019-09-03 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-01

CONDITIONS: Pharmacology

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HM15912 (Experimental)
  Interventions: Drug: HM15912
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: HM15912 — The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
  Arms: HM15912
Drug: Placebo — The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
  Arms: Placebo

SUMMARY:
A First-in-Human, Double-blind, Randomized, Placebo-controlled, Single Ascending Dose Study to Assess Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of HM15912 in Healthy Korean Subjects

ELIGIBILITY:
Inclusion Criteria:

* Subject voluntarily agrees to participate in this study and signs an IRB-approved informed consent prior to performing any of the Screening visit procedures.
* Korean males and females ≥ 19 and ≤ 60 years of age at the Screening visit

Exclusion Criteria:

* Subject with a history or presence of clinically significant active diseases.
* Subject who has participated in other clinical studies (including bioequivalence tests) within 6 months before the Screening visit and has received IPs

Ages: 19 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-10-08 (Actual); Primary Completion 2020-11-10 (Actual); Study Completion 2021-05-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Date of first enrollment was October 8th, 2019.
Pre-assignment Details: The planned maximum dose of HM15912 was 1.5 mg/kg; however, higher doses were allowed to be administered if safety was confirmed in previous cohorts. If dose was escalated to more than 1.5 mg/kg, Ministry of Food and Drug Safety (MFDS) approval was to be obtained.
Groups:
- HM15912 0.05mg/kg; HM15912 0.1mg/kg; HM15912 0.5mg/kg; HM15912 1.0mg/kg; HM15912 1.5mg/kg: HM15912: The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
- Placebo: Placebo: Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo). Total of 10 subjects for placebo.
Period: Overall Study
Arm/Group | HM15912 0.05mg/kg | HM15912 0.1mg/kg | HM15912 0.5mg/kg | HM15912 1.0mg/kg | HM15912 1.5mg/kg | Placebo
Started | 6 | 6 | 6 | 6 | 6 | 10
Completed | 6 | 6 | 6 | 6 | 6 | 10
Not Completed | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- HM15912 1.0 mg/kg; HM15912 1.5mg/kg: HM15912: The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
- Total: Total of all reporting groups
Arm/Group | HM15912 0.05mg/kg | HM15912 0.1mg/kg | HM15912 0.5mg/kg | HM15912 1.0 mg/kg | HM15912 1.5mg/kg | Placebo | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 40
Age, Continuous [Mean (Standard Deviation); unit: Years] | 31 (5.18) | 28.3 (8.87) | 26.0 (5.83) | 25.0 (3.52) | 31.7 (7.39) | 27.2 (2.39) | 28.4 (6.54)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Male | 6 | 6 | 6 | 6 | 6 | 10 | 40
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Korean | 6 | 6 | 6 | 6 | 6 | 10 | 40
Region of Enrollment [Number; unit: participants]
  South Korea | 6 | 6 | 6 | 6 | 6 | 10 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-emergent Adverse Events of HM15912
Description: Number of participants with any treatment-emergent adverse events related to study medication.
Time Frame: after single subcutaneous (SC) doses for 44 days
Population: Each analysis population was included in the analyses, based on the actually administered IMP and dosage.
Measure: Count of Participants; unit: Participants
Arm/Group | HM15912 0.05mg/kg | HM15912 0.1mg/kg | HM15912 0.5mg/kg | HM15912 1.0mg/kg | HM15912 1.5mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants
  Mild TEAE | 3 | 1 | 2 | 4 | 4 | 5
  Moderate TEAE | 0 | 2 | 0 | 0 | 0 | 1
  No AE | 3 | 3 | 4 | 2 | 2 | 4

2. Primary Outcome: Number of Participants With Significant Findings Observed for Hematology
Time Frame: after single subcutaneous (SC) doses for 44 days
Measure: Count of Participants; unit: Participants
Arm/Group | HM15912 0.05mg/kg | HM15912 0.1mg/kg | HM15912 0.5mg/kg | HM15912 1.0mg/kg | HM15912 1.5mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
Participants | 0 | 0 | 0 | 0 | 0 | 0

3. Secondary Outcome: Concentration Max Profile of HM15912
Description: To assess the Concentration Max profile of HM15912 after single SC doses.
Time Frame: after single subcutaneous (SC) doses at day 1,2,3,4,5,6,7,10,17 and 30
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | HM15912 0.05mg/kg | HM15912 0.1mg/kg | HM15912 0.5mg/kg | HM15912 1.0mg/kg | HM15912 1.5mg/kg | Placebo
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10
ng/mL | 249.45 (51.77) | 622.46 (14.06) | 3550.79 (36.44) | 8347.70 (10.30) | 9393.06 (13.24) | 0 (0)

ADVERSE EVENTS:
Time Frame: Screening, Day1 to 7, Day 10, Day 17, and Day 30
Description: An AE was defined as any untoward medical occurrence in subjects and which did not necessarily have a causal relationship with the IMP. An AE could therefore have been any unfavorable and unintended sign (including abnormal laboratory findings), symptom or disease, whether or not it was related to the IP.
Groups:
- HM15912 0.05mg/kg: HM15912 0.05mg/kg: The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
- HM15912 0.1mg/kg: HM15912 0.1mg/kg: The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
- HM15912 0.5mg/kg: HM15912 0.5mg/kg: The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
- HM15912 1.0mg/kg: HM15912 1.0mg/kg: The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
- HM15912 1.5mg/kg: HM15912 1.5mg/kg: The study will be conducted in approximately 5 sequential dosing cohorts, enrolling 8 subjects per cohort. Subjects will be randomized to HM15912 or placebo in a ratio of 6:2 (6 active, 2 placebo).
Arm/Group | HM15912 0.05mg/kg | HM15912 0.1mg/kg | HM15912 0.5mg/kg | HM15912 1.0mg/kg | HM15912 1.5mg/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10
Other Adverse Events (participants affected / at risk) | 3/6 | 3/6 | 2/6 | 4/6 | 4/6 | 6/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HM15912 0.05mg/kg (N=6) | HM15912 0.1mg/kg (N=6) | HM15912 0.5mg/kg (N=6) | HM15912 1.0mg/kg (N=6) | HM15912 1.5mg/kg (N=6) | Placebo (N=10)
Injection site bruising (General disorders) | 0 | 0 | 0 | 2 | 3 | 2
Headache (Nervous system disorders) | 2 | 0 | 0 | 0 | 1 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2 | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 0 | 1 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-04-06): https://cdn.clinicaltrials.gov/large-docs/93/NCT04076293/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-18): https://cdn.clinicaltrials.gov/large-docs/93/NCT04076293/SAP_001.pdf